CLINICAL TRIAL: NCT07187466
Title: Sequential Multiple Assignment Randomized Trial to Treat Urinary Symptoms in Parkinson Disease
Brief Title: Behavioral and/or Mirabegron to Treat Urinary Symptoms in Parkinson Disease
Acronym: SQUARE PD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RRD6-001-24W
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder; Parkinson Disease
Keywords: Urinary Bladder, Overactive; Parkinson Disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Parkinson Disease | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART) design offers an efficient strategy to understand both intervention and patient factors that will inform an individualized treatment plan. With a SMART design, Aim 1 will determine if non-responders to behavioral or drug treatment (expected to be 50% of population) demonstrate a clinically significant response to combination behavior and drug treatment compared to a single treatment approach. In Aim 2, the investigators will determine patient factors that influence optimized treatment of urinary symptoms in Veterans with PD.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Drug Therapy Group (Active Comparator): Participants who are randomized to drug therapy will receive mirabegron 25mg at visit 2 (randomization visit).
  Interventions: Drug: mirabegron
- Behavioral Therapy Group (Active Comparator): Participants who are randomized to exercise-based behavioral therapy will receive a comprehensive training program administered individually by a trained nurse practitioner interventionist to address urinary incontinence and other lower urinary tract symptoms.
  Interventions: Behavioral: Exercise-based behavioral therapy
- Combined Drug and Behavioral Therapy Group (Active Comparator): At 6 weeks post-randomization, participants will complete the ICIQ-OAB questionnaire. Participants reporting less than 2 points reduction will be re-randomized to either continue their initial treatment assignment or receive combination therapy by adding the alternate treatment strategy, thus participants initially treated with mirabegron will add behavioral therapy and participants initially treated with behavioral therapy will add mirabegron.
  Interventions: Drug: mirabegron; Behavioral: Exercise-based behavioral therapy

INTERVENTIONS:
Drug: mirabegron — Mirabegron is a beta-3-agonist, which acts upon the noradrenergic system and avoids the cognitive and gastrointestinal side effects of anticholinergic bladder relaxants.
  Other Names: Myrbetriq
  Arms: Combined Drug and Behavioral Therapy Group; Drug Therapy Group
Behavioral: Exercise-based behavioral therapy — The exercise-based behavioral therapy is a comprehensive training program administered individually by a trained nurse practitioner interventionist to address urinary incontinence and other lower urinary tract symptoms.
  Arms: Behavioral Therapy Group; Combined Drug and Behavioral Therapy Group

SUMMARY:
The purpose of this study is to learn about different treatments for overactive bladder symptoms in Parkinson's Disease. The investigators want to find out if people who do not respond to one treatment (either behavioral or drug treatment) will respond to combined treatment. The investigators also want to find out what factors influence whether someone responds to the treatments.

DETAILED DESCRIPTION:
While PD is often characterized by the motor symptoms of the disease (tremor, bradykinesia, rigidity), non-motor symptoms such as urinary symptoms correlate more closely with impaired well-being as the disease progresses. The urinary symptoms of overactive bladder (OAB), including urgency, frequency, and nocturia, with or without urinary incontinence, are the most common urinary symptoms of PD. Because OAB symptoms, such as incontinence and nocturia, are associated with falls (a cause of increased mortality in PD), spouse/caregiver stress, and, ultimately institutionalization, it is critical that the investigators optimize the care of urinary symptoms for Veterans with PD. In the non-PD population, pelvic floor muscle contractions diminish bladder muscle contraction and recent evidence demonstrates that behavioral training with pelvic floor muscle exercises improves the cortical integration of bladder afferent signals. Because of its effectiveness compared to drugs, pelvic floor muscle exercise-based behavioral therapy is recommended first-line in men and women without PD who have OAB. Pelvic floor muscle exercise-based behavioral therapy for urinary symptoms requires individuals to learn a motor skill and implement an adaptive behavioral strategy incorporating pelvic floor muscle contraction to delay the need to void when urgency strikes. The PI's research group demonstrated the feasibility and preliminary efficacy of pelvic floor muscle exercise-based behavioral therapy to treat urgency incontinence in adults with PD. However, the most recent clinical guidelines for the treatment of urinary symptoms in PD recommend treatment with anticholinergic drugs and mention the potential option for noradrenergic bladder relaxants. While some anticholinergic drugs are effective in reducing symptoms of OAB, it is important to note that there is a glaring lack of an empirical evidence base to promote these drugs in the setting of PD given that they add to the anticholinergic burden of antiparkinsonian therapy and may worsen the cognitive and autonomic burdens of the illness. Noradrenergic bladder relaxants may have a more favorable side effect profile; however, the evidence for efficacy in PD is minimal. Therefore, randomized controlled trials (RCTs) are needed to optimize treatment paradigms for urinary symptoms in PD. The investigators' preliminary studies suggest adults with PD and mild cognitive dysfunction can successfully implement behavioral therapy for urinary symptoms. However, in the investigators' most recent VA-funded, multisite trial, 50% of participants reported a clinically significant reduction in urinary symptoms after treatment with either behavioral or drug treatment. Additional research using a Sequential Multiple Assignment Randomized Trial (SMART) design offers an efficient strategy to understand both intervention and patient factors that will inform an individualized treatment plan. With a SMART design, Aim 1 will determine if non-responders to behavioral or drug treatment (expected to be 50% of population) demonstrate a clinically significant response to combination behavior and drug treatment compared to a single treatment approach. In Aim 2, the investigators will determine patient factors that influence optimized treatment of urinary symptoms in Veterans with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD determined by a board-certified neurologist with specialty training in movement disorders
* An ICIQ-OAB Symptom Score of 7 or higher, which indicates clinically significant symptoms of OAB, defined as presence of urinary urgency with or without urgency incontinence usually with increased daytime frequency and nocturia in the absence of infection or other obvious pathology

Exclusion Criteria:

* Significant cognitive impairment, as indicated by a Montreal Cognitive Assessment (MoCA) score of < 18 or a telephone-MoCA score < 13, which is the recommended diagnostic cut point for dementia in PD.
* Previous intensive pelvic floor muscle exercise training
* Clinically significant depression as measured by a Geriatric Depression Scale-Short Form score of 10 or higher which could affect motivation to fully engage in the intervention
* Use of an indwelling urinary catheter
* Post-void residual urine measurement by bladder ultrasound of > 150 mL
* Severe uterine prolapse past the vaginal introitus
* Poorly controlled diabetes defined by a hemoglobin A1c (HgbA1c) of >9.0% within the last 3 months. Participants with poorly controlled diabetes will be offered enrollment if the OAB symptoms persist after improvement in diabetes control
* Chronic renal failure and on hemodialysis
* Genitourinary cancer with ongoing surgical or external beam radiation treatment
* Previous artificial urinary sphincter, sling procedure or implanted sacral neuromodulation device
* History of bladder-injection of botulinum toxin in the last 12 months
* Any unstable health condition expected to result in hospitalization or death within in the next 3 months as determined by principal investigator.
* Hypersensitivity to drug class
* Contraindication to the study drug (mirabegron) including history of acute urinary retention requiring catheterization
* Current use of a bladder relaxant - permitted to enroll after one-week washout
* Hematuria on microscopic examination in the absence of infection. A urologic consultation will be recommended, and enrollment will depend on clearance by a urologist and agreement by the site PI that entry into the treatment protocol is not contraindicated
* If on diuretic, dose should be stable for at least 4 weeks
* If taking an alpha-blocker, dose should be stable for at least 4 weeks
* If taking dutasteride or finasteride, dose should be stable for at least 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
ICIQ-OAB | baseline, 6-weeks, and 12-weeks
  The primary outcome measure at 12 weeks will be urinary symptom severity as measured by the International Consultation on Incontinence Questionnaire-Overactive Bladder module (ICIQ-OAB). Scores range from 0 to 16 with higher scores indicating worse symptom frequency. The symptom score will be collected at 3 time points during the study: baseline, 6-weeks, and 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Camille Vaughan, MD MS, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying publications resulting from the proposed research will be shared outside VA through a de-identified, anonymized Dataset under a written agreement that adheres to any applicable Informed Consent provisions and prohibits the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.